CLINICAL TRIAL: NCT03792048
Title: Magnetic Compressive Anastomosis for Biliojejunostomy and Pancreaticojejunostomy During Whipple's Procedure: a Prospective Case-control Study
Brief Title: Magnetic Compressive Anastomosis for Biliojejunostomy and Pancreaticojejunostomy During Whipple's Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-001-2
Record Dates: First submitted 2018-12-12; First posted 2019-01-03 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Cholangiocarcinoma; Pancreatic Neoplasms; Duodenal Neoplasms; Pancreatolithiasis; Chronic Pancreatitis
Keywords: bilioenteric anastomosis; pancreaticojejunostomy; Magnetic Compressive
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Duodenal Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Compressive Anastomosis (Experimental): A magnetic device will be used during bilioenteric anastomosis and pancreaticojejunostomy
  Interventions: Procedure: Magnetic Compressive Anastomosis
- Manual Anastomosis (No Intervention): Manual Anastomosis for bilioenteric anastomosis and pancreaticojejunostomy

INTERVENTIONS:
Procedure: Magnetic Compressive Anastomosis — A magnetic device will be used during bilioenteric anastomosis and pancreaticojejunostomy
  Arms: Magnetic Compressive Anastomosis

SUMMARY:
Magnetic anastomosis has been attempted in biliary and intestinal reconstruction. Based on our initial experience, the investigators have successfully utilized magnetic anastomosis for biliojejunostomy and pancreaticojejunostomy during pancreaticoduodenectomy. The current study was to design a prospective and case-control study with utilization of magnetic compression anastomosis for pancreaticojejunostomy and biliojejunostomy in Whipple's procedure versus traditional hand-sewn technique on the postoperative morbidity, such as biliary/pancreatic fistula, hemorrhage, anastomotic stenosis, etc. In addition, the investigators are seeking to assess the safety and formation of the anastomosis by magnetic technique.

DETAILED DESCRIPTION:
The magnets used in the current study consists of a mother and daughter magnets. An 8-Fr nasogastric tube is tightly fixed with the mother magnet, which will be used for bile or pancreatic drainage before formation of anastomoses. The outside diameter (OD) of the magnets ranges from 5mm to 15mm. In fact, for biliojejunostomy, larger magnets are applied, whereas for pancreaticojejunostomy, smaller magnets are routinely used. This study is a single-center, parallel controlled trial to evaluate the safety and effectiveness of magnetic compression technique for biliojejunostomy and pancreaticojejunostomy, versus traditional hand-sewn techniques on the postoperative morbidity of the patients. And also how to avoid mutual attraction of the two pairs of magnets, formation of bilio-/pancreaticojejunostomy time, discharge rule of the magnets will be all evaluated in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 to 75
* Patients' gender was not limited
* Patients who were well-diagnosed and had the indication for anastomosis.
* Patients whose lifetimes will be longer than 12 months.
* Patients who are willing to join this clinical trial and informed consent form voluntarily.

Exclusion Criteria:

* Woman during pregnancy or lactation or anyone with mental disorder
* The wall of biliary duct or jejunum was too thick so that the attractive force of magnetic device cannot meet the requirements of compression.
* Any anatomical variation in bile ducts system or the inner diameter is too small so that the magnetic device cannot place in.
* Any foreign body has been implanted in body, such as heart pacemaker.
* Surgical contraindication, including:

Child-Pugh C with hepatic encephalopathy Anyone with heart, lung, kidney dysfunction or other organ dysfunction, and cannot tolerate surgery.Hepatic ducts stone disease, who was diagnosed as Acute Cholangitis of Severe Type, especially complicated with bacteremia or septic shock. End stage disease, complicated with biliary cirrhosis or portal hypertension.Patients with long-term obstructive jaundice, dehydration, electrolyte disturbance or coagulation defects; Patients have the tendency or history of bleeding.

-Any other disease in perioperation periods which needs MRI examination in the next 8 weeks post operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of anastomotic fistula | 1 month post operation
  Incidence of biliary or pancreatic fistula after surgery

SECONDARY OUTCOMES:
Length of bilio-/pancreaticojejunostomy time | during operation
  Separate operation time of magnetic anastomosis for bilio- and pancreaticojejunostomy
average length of postoperative hospital stay | 1 to 4 weeks postoperation
  length of hospital stay (days) after surgery
Hospitalization cost | 1 to 4 weeks postoperation
  cost in hospital
incidence of biliojejunostomic stricture | 12 months post operation
  Incidence of biliojejunostomic stricture between magnetic and manual groups during the relatively long-term follow-up
Incidence of pancreaticojejunostomic stricture | 12 months post operation
  Incidence of pancreaticojejunostomic stricture between magnetic and manual groups during the relatively long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided